CLINICAL TRIAL: NCT04286464
Title: Early Environmental and Maternal Determinants of Airway Inflammation in Wheezing Disorders in Infants
Status: Enrolling by invitation | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BILD
Record Dates: First submitted 2019-10-09; First posted 2020-02-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers
Keywords: infants; children; healthy; term born; preterm born; fetal growth restriction; intrauterine growth restriction or preeclampsia; with gestational diabetes; with IVF or amnion dysfunction
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs, oropharyngeal swabs, nasal brush, sputum, cord blood, blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Term born group (H): Healthy, white and term Born infants and Children Born 38-42 weeks postconceptional
  Interventions: Other: No intervention
- Preterm group (P): Healthy, white preterm Born infants and Children Born <37 weeks postconceptional Which comply with the international criteria (Jobe and Bancalari) of a diagnosis of bronchopulmonary dysplasia (BPD), or of chronic lung disease of the new-born (CLD)
  Interventions: Other: No intervention
- Risk pregnancy group (RP): White preterm Born infants and Children, including Twins Born <37 weeks postconceptional With fetal growth restriction (FGR), intrauterine growth restriction (IUGR) or preeclampsia (PE) With gestational Diabetes (GDM) With IVF or Amnion dysfunction
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study collects data on microbiological, genetic and environmental factors, as well as lung function parameters (e.g. spirometry, body plethysmography, lung-MRI) to assess the complex interaction of predisposing risk factors for impaired lung development and respiratory diseases.

DETAILED DESCRIPTION:
Background:

Lung development and growth is a complexly orchestrated process starting prenatally in the first embryonic weeks, and ending, with the last important stages of alveolarization from the 24th week onwards. By the time of birth, around one third of the total amount of alveoli has developed, while the rest develops during infancy and childhood. After birth, lung volume, airways and the gas-exchanging surface increase by a multiple, reaching the maximum lung size at around 25 years of age. A comprehensive understanding of lung growth and development is crucial in order to understand the pathophysiology of lung diseases. During childhood and ongoing lung growth, an important amount of respiratory diseases might develop.

Objectives:

Longitudinal assessment of lung growth and development, to examine respiratory morbidity such as Asthma and allergy, and the complex relationship between associated Risk factors mainly genetic predisposition and environmental factors on both lung development and subsequent respiratory morbidity, Therefore, longitudinal data on lung function and structure, on respiratory morbidity and on genetic, immunological, microbiological and environmental risk factors will be collected.

Methods:

Recruitment and participation:

Participants will be recruited antenatal through advertisement placed at gynaecological Hospital in Bern and by obstetricians or midwives. Interested participants can get further information about the study by telephone from study nurses, as well as during the baseline visit at the University Children's Hospital in Bern, respectively. Mothers with a high risk of a preterm delivery will be informed by clinical Investigators at the Department of Obstetrics of the University Hospital Bern. Preterm infants, which receive ventilatory support over a long period are at Risk for chronical lung diseases in early childhood, named bronchopulmonary dysplasia (BPD). The recruitment of this infants will take place at the neonatology intensive care unit by clinical Investigators. On average 40 healthy children, 40 preterm children and 20 infants from risk pregnancies will be recruited as participants of the BILD cohort each year for Study Phase I. At 3, 6, 9, 12, 15 years and once after the 16th year of age the parents/participants will be asked again, if they would like to participate at the follow-up visits at the University Children's Hospital in Bern for the subsequent Study Phases II and III.

Information collected:

Lung function data:

* Tidal breathing parameters (minute ventilation, respiratory rate, tidal volume, tidal expiratory flow, tidal inspiratory flow, time to peak expiratory flow) averaged over 100 breaths.
* Multiple breath washout (FRC, LCI, moment ratios) and single breath washout (molar mass)
* Fractional exhaled nitric oxide (marker of airway inflammation)
* Spirometric forced expiratory volume loops (FVC, FEV1, PEF, MEF50)
* Body plethysmography (airway resistance, lung volumes: TLC, FRC, RV)
* Respiratory Rate over 60 seconds
* Interrupter resistance measurement (RINT)
* Volatile organic compounds
* Forced oscillation technique (FOT)
* Electrical impedance tomography (EIT)
* Impedance plethysmography (IP)

Microbiological data:

* Nasal swabs (respiratory virus and bacterial diagnostics, as well as host transcriptome Analysis)
* Pharyngeal swabs (bacterial colonization and microbiota Analysis)
* Anterior nasal and oropharyngeal swabs (viral, bacterial and host transcriptome Analysis)
* Nasal brush
* Sputum (to analyse the neutrophils)

Cord blood (mononuclear cells (CBMC) (e.g. lymphocytes)which regulate the innate and adaptive immunity)

Blood count (hemoglobin concentration, hematocrit, leukocyte number, lymphocyte number, lymphocyte count, eosinophil count, basophil count, monocyte count, promyelocyte count, myelocyte count, platelet count, immunoglobulin E Level, Interleukins, Granulocyte-Monocyte-Colony Forming Unit, Tumor Necrosis Factor alpha, Interferon gamma and Interferon lambda)

Urin (to estimate the tobacco exposure during pregnancy (amount of Cotinine) and the content of caffeine and Steroid profile)

Lung function MRI: functional and structural images of the lung

Environmental pollution (Level of particulate matter <10um, Nitrogen dioxide, ozone and particulate matter <2.5um)

Skin-Prick Test (test for pollen, trees, house dust mite, cat and dog)

Questionnaires (to assess quality of life)

Medical history (information on respiratory Symptoms, pulmonary exacerbations, hospitalisations and regular therapy)

Study database:

All study data is recorded in an Access-database with SQL Servers by electronic Case Report Forms. The database is accordant to the HFG and was adapted together with the CTU.

Funding:

Schweizerischer Nationalfonds (SNF) and Departement Lehre und Forschung of the Inselspital Bern.

ELIGIBILITY:
Inclusion Criteria:

* Term Born group (H): Healthy, white and term Born infants and Children. Born 38-42 weeks postconceptional.
* Preterm group (P): Healthy, white preterm Born infants and Children. Born <37 weeks postconceptional. Which comply with the international criteria (Jobe and Bancalari) of a diagnosis of bronchopulmonary dysplasia (BPD), or of chronic lung disease of the new-born (CLD).
* Risk pregnancy group (RP): White preterm Born infants and Children, including Twins. Born <37 weeks postconceptional. With fetal growth restriction (FGR), intrauterine growth restriction (IUGR) or preeclampsia (PE). With gestational Diabetes (GMD). With IVF or Amnion dysfunction.
* Parents: language skills in German or French (by at least one parent).
* Both of the parents can be Smokers and may be atopics (allergy of the mother and/or the Father).
* Signed, written informed consent of the parents.

Exclusion Criteria:

* Term Born group (H): Need of respiratory support > three days postnatal. Severe malformations or known diseases. Maternal drug abuse except smoking. Known sever maternal disease postpartum. Insufficient Knowledge of Project language (no German or French speaker). Pacemaker, continuous glucose monitor.
* Preterm group (P): Severe malformations or known diseases. Maternal drug abuse except smoking. Known severe maternal disease postpartum. Insufficient Knowledge of Project language (no German or French speaker). Pacemaker, continuous glucose monitor.
* Risk pregnancy group (RP): Insufficient Knowledge of Project language (no German or French speaker). Concurrent participation in another study. Participants, which lead to heterogeneity in genetic analysis and thus preclude any findings.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healty term born, healthy preterm born infants and children and white preterm born infants and children from risk pregnancies.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2003-09 (Actual); Primary Completion 2050-09 (Estimated); Study Completion 2051-01 (Estimated)

PRIMARY OUTCOMES:
Change in Multiple Breath Washout | Every third year from the age of 4-6 weeks/1 year till >16 years.
  Longitudinal assessment of lung volume and ventilation inhomogeneity
Change in Spirometry | Every third year from the age of 4-6 weeks/1 year till >16 years
  Longitudinal assessment of long volumes
Change in Body plethysmography | Every third year from the age of 4-6 weeks/1 year till >16 years.
  Longitudinal assessment of ventilation inhomogeneity.
Change in Magnetic Resonance Imaging (MRI) | At the age of 4-6 weeks, 1, 3, 6, 9, 12, 15 and >16 years.
  Longitudinal assessment of regional lung perfusion and ventilation
Change in Nasal swabs | At the age of 4-6 weeks, 1, 3, 6, 9, 12, 15 and >16 years.
  Longitudinal assessment of viral and bacterial colonization of the nasal swab
Change in Weekly swabs | Weekly from the visit at the age of 8-12 weeks till the age of 1 year.
  Respiratory virus and bacterial diagnostic
Swabs during respiratory infection | Any timepoint between the visit at the age of 4-6 weeks till the age of 1 year.
  Respiratory viruses and Bacteria, changes of the microbial flora

SECONDARY OUTCOMES:
Respiratory Rate (RR) | From the visit at the age of 4-6 weeks till the age of 1 year.
  The number of breaths over 60 seconds
Urine | At the age of 4-6 weeks.
  Estimation of tobacco exposure during pregnancy.
Cord blood | At birth.
  Assessment of mononuclear cells, which regulate the innate and adaptive immunity.
Capillary blood markers | At the age of 1, 3, 6, 9, 12, 15 and >16 years.
  Assessment of blood markers.
Skin Prick Test | At the age of 3, 6, 9, 12, 15 and >16 years.
  Assessment of the history of atopy and allergy
Environmental pollution markers | At the age of 4-6 weeks, 1, 3, 6, 9, 12, 15 and >16 years.
  Level of particulate matter <10um, Nitrogen dioxide, ozone and particulate matter <2.5um.
Volatile organic compound markers | At the age of 4-6 weeks, 1, 3, 6, 9, 12, 15 and >16 years.
  Real-time Analysis of gases.
Oropharyngeal swabs | At the age of 1, 3, 6, 9, 12, 15 and >16 years.
  Longitudinal assessment of viral and bacterial colonization.
Nasal brushes | At the age of 1, 3, 6, 9, 12, 15 and >16 years.
  Longitudinal assessment of viral and bacterial colonization.
Sputum | At the age of (3), 6, 9, 12, 15 and >16 years.
  Longitudinal assessment of the sputum neutrophils.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Latzin, MD PhD, Principal Investigator — University Children's Hospital Bern
Locations (1):
- University Children's Hospital, Bern, Switzerland